CLINICAL TRIAL: NCT02987153
Title: Kypho-Intra Operative Radiation Therapy (IORT) for Localized Spine Metastasis, Phase I/II Study
Acronym: Kypho-IORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Maged Ghaly, Asst. Professor of Radiation Medicine, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-298
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Spinal Metastases
Keywords: Kyphoplasty; Spinal metastases; IORT; Intraoperative radiation therapy; Pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KYPHO-IORT - 10 Gy and Kyphoplasty (Experimental): Intra-operative radiation therapy followed by standard kyphoplasty
  Interventions: Radiation: Kypho-IORT

INTERVENTIONS:
Radiation: Kypho-IORT — The radiation source is inserted into the lesion and switched on for a few minutes to provide intraoperative radiotherapy accurately targeted to the tissues that are at the highest risk of local recurrence. The dosimetric characteristics and clinical applications of this device have been well studied.
  Other Names: Intrabeam® Photon Radiosurgery System

SUMMARY:
Kypho-IORT is a novel approach to combine kyphoplasty, a minimally invasive procedure, with a single dose of intraoperative radiotherapy (IORT) for the treatment of unstable or potentially unstable spinal cord metastases. The primary objective is to evaluate the response rate of pain control when combining kyphoplasty, a minimally invasive procedure, with a single dose of intraoperative radio- therapy (IORT) for the treatment of spinal cord metastases. Secondary objectives are (i.) to determine feasibility for unstable or potential unstable spine metastases; (ii.) to determine tolerability/side effects of the IORT within 90 days post-procedure; (iii.) to determine which clinical factors are prognostic of vertebral compression fracture

DETAILED DESCRIPTION:
Approximately 20% of patients with spine metastasis present with unstable lesions, which represent a common therapeutic dilemma in patients with advanced stage cancer and limited survival time. Management necessitates spinal stabilization surgery such as laminectomy, vertebroplasty, or kyphoplasty for mechanical back pain control and irradiation for the underlying malignant process. Because of the limited survival time of patients with metastatic cancer, novel, more convenient treatment concepts to shorten the overall treatment time or hospitalization are desirable. We developed a novel approach to combine kyphoplasty, a minimally invasive procedure, with a single dose of intraoperative radio- therapy (IORT) for the treatment of spinal cord metastases.

Patients treated with Kypho-IORT will receive a prescribed dose of 8 Gy in 1 fraction from The Intrabeam® Photon Radiosurgery System source. The target volume includes only the tumor. The technique of the operation and the delivery of radiotherapy has been described and published previously. TARGiT Academy training and requisite test cases have been completed prior to enrolling subjects on this study. The balloon kyphoplasty, which is an advancement of the vertebroplasty, is a treatment option for fractured vertebral bodies which utilizes bone cement to provide needed support.

Outcome measures will include complete or partial pain relief or a stable response at the index site requiring no increase in narcotic pain medication. Therefore, patients with complete or partial pain relief will be considered responders. Patients with complete or partial pain relief at the index site but a progressive response at the secondary site(s) will be considered non-responders.

Quality of Life Measurements. It is hypothesized that quality of life (QOL) will improve after Kypho-IORT due to rapid and durable pain control after spine treatment. In the current study, we will measure the QOL [EORTC QLQ-C30 (version 3)], the Brief Pain Inventory (BPI), ambulation , and steroid and narcotic use pre- and post-procedure at 1-week, 3-month, 6-month, 9-month, 1-year, and 2-year intervals. The involved spine will be imaged at 3-month intervals up to one year, and at 2 years post-procedure.

All the evidence to date supports the description of the Intrabeam as delivering an accurate and reliable dose. Physicists on site will be responsible for verifying the miniature x-ray source is operational prior to use and setting up the parameters within the control console software for treatment delivery. During the procedure, the control console monitors the system for safe and accurate dose delivery.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky Index ≥ 60.
* History/physical examination within 4 weeks prior to procedure.
* Imaging of the involved spine within 8 weeks prior to procedure to determine the extent of the spine involvement.
* Numerical Rating Pain Scale within 4 week prior to procedure (score must be ≥ 5 for at least one of the planned sites for spinal IORT.
* Neurological examination within 4 week prior to procedure to rule out rapid neurologic decline.
* Spine Instability Neoplastic Score (SINS score) = ≤12.
* Negative serum pregnancy test within 4 weeks prior to procedure for women of childbearing potential.
* Women of childbearing potential and male participants who are sexually active must agree to use a medically effective means of birth control.
* The patient must have localized spine metastasis from the T5 to L5 levels by a screening imaging study [bone scan, PET, CT, or MRI] (a solitary spine metastasis; two separate spine levels; or up to 3 separate sites are permitted). Each of the separate sites have a maximal involvement of ONE vertebral body. Patients can have other visceral metastasis.
* Patients must provide study specific informed consent prior to study entry.

Exclusion Criteria:

* Spine instability due to a compression fracture; SINS score >12.
* Frank spinal cord compression or displacement or epidural compression within 3 mm of the spinal cord
* Patients with rapid neurologic decline
* Bony retropulsion causing neurologic abnormality
* Patients allergic to contrast dye used in MRIs or CT scans or who cannot be premedicated for the use of contrast dye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-11; Primary Completion 2022-07 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
To evaluate pain control | 90 days
  To evaluate the response rate of pain control when combining kyphoplasty, a minimally invasive procedure, with a single dose of intraoperative radio- therapy (IORT) for the treatment of spinal cord metastases.

SECONDARY OUTCOMES:
Feasibility of Kypho-IORT as treatment modality | 90 days
  To determine the feasibility of delivered Kypho-IORT for unstable or potential unstable spine metastases.
Tolerability/side effects | 90 days
  To determine tolerability/side effects of the IORT based on defined MTD criteria (wound healing problems, infection, osteoradionecrosis, nerve and spinal cord damage, pathological fracture, secondary fractures/sintering progression and symptomatic or asymptomatic cement leakage within 90 days.
Local tumor control | 2 years
  Local tumor control is defined as no recurrent tumor in the treated lesion. Patients will be regularly monitored as per the site's policy provided this meets the minimum trial criteria for follow-up with physical examination 1 week post treatment, and at 3 months, 6 months, 1 year, and 2 years post-treatment.
Overall survival | 2 years
  Overall survival will be the time interval between enrollment and death.
Measures of quality of life. | 2 years
  Evaluate the potential benefit of Kypho-IORT on change in and overall quality of life, in pain as measured by the Brief Pain Inventory (BPI); Ambulation, and EORTC QLQ-C30 (version 3).
Steroid and narcotic use. | 2 years
  The average daily morphine equivalent (mgs) used.

CONTACTS AND LOCATIONS:
Overall Officials: Maged Ghaly, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health, Lake Success, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data